CLINICAL TRIAL: NCT01639027
Title: Use of Antispasmodic Drotaverine to Shorten the Length of Labor in Nulliparous Women
Brief Title: Drotaverine to Shorten the Length of Labor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohammed Abd El Hameed Abd El Lateef, Investigator, Obstetrics and Gynaecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Drotaverine in labor
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Prolonged First Stage of Labor; Failure of Cervical Dilation as Antepartum Condition; Labor Pain; Mild Birth Asphyxia, APGAR 4-7
MeSH Terms: conditions — Labor Pain | interventions — drotaverin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drotaverine (Active Comparator): Women who will receive 40 mg Drotaverine hydrochloride (Do-Spa) IV injection.
  Interventions: Drug: Drotaverine
- Placebo (Placebo Comparator): Women who will receive 2ml of normal physiological saline (0.9% sodium chloride) I.V.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drotaverine — 40 mg Drotaverine hydrochloride (Do-Spa) IV injection at the start of the study and repeated every 2 hours up to a maximum 3 injections.
  Other Names: Do Spa
  Arms: Drotaverine
Drug: Placebo — Women who will receive 2ml of normal physiological saline (0.9% sodium chloride) I.V at the start of the active phase of labor.
  Other Names: Normal physiological saline (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
Reducing the length of labor is a highly desirable goal of intrapartum care, both from a perspective of maternal and fetal well-being, and for the providers of the birth services. Avoiding along, protracted labor entails shorter exposure to pain, anxiety and stress and would thus translate into a major improvement in maternal satisfaction with the childbirth experience.

Based on the premise that shortening the length of labor is beneficial, interventions aimed at accelerating the progression of labor have been introduced routinely as part of standard labor management and care throughout the 20th century. Certain labor accelerative procedures, such as amniotomy, became common practice and have been put to the acid test of randomized control trials to evaluate their efficacy. Use of anticholinergics/antispasmodics as a method of augmenting labor was ﬁrst described in 1937 by Hirsch, who reported a decrease in labor length by two to four hours following Intrapartum administration of an atropine-like drug (Syntropan®)mainly among older nulliparas.

Drotaverine, an isoquinolone derivative is a superior smooth muscle relaxant which acts specifically on spastic sites and corrects the cAMP and calcium balance relieving smooth muscle spasm.

This inhibitory action is detected only in lower uterine segment during labor since muscle fibers in upper uterine segment are strongly affected by contractile effect of oxytocin. Use of drotaverine during pregnancy is free of any teratogenic and embryotoxic effects.

The Research question is: Does the use of antispasmodic Drotaverine shorten the duration of active first stage of labor in nulliparous women as compared to placebo?

DETAILED DESCRIPTION:
Research question:

Does the use of antispasmodic Drotaverine shorten the duration of active first stage of labor in nulliparous women as compared to placebo?

Research hypothesis: the population means of the Drotaverine and placebo groups are equal regarding the duration of the first stage of labor.

Objectives:

The purpose of this study was to determine the effectiveness of Drotaverine for reducing the duration of labor for the context of contemporary practice, among nulliparous women managed according to a standard intrapartum protocol.

Study setting:

Patients will be recruited from women admitted in labor at the delivery unit of Ain Shams Maternity Hospital.

Study design:

This study is a phase II to III, intervention study- Randomized Controlled double blind study.

Procedure:

Every patient will be subjected to:

1. Complete history to exclude allergy to Drotaverine Hydrochloride and any contraindication for normal vaginal delivery.
2. General examination of the patients including (pulse, blood pressure, temperature).
3. Obstetric Abdominal examination including lie, presentation,station; fetal heart rate, uterine contraction, amount of liquor and to exclude multiple pregnancies.
4. Vaginal examination under aseptic conditions to assess cervical dilation, effacement, state of fetal membranes, presenting part,position of fetal head, color of liquor and pelvic adequacy.
5. Assessment of the frequency, duration of uterine contractions and monitoring of fetal wellbeing will be applied through CTG application on admission:

   - CTG will be applied half an hour to all participants before starting any intervention.
   1. If the contractions are not adequate:

      * Patients with intact membranes → AROM will be done, reassessment after one hour. If still no adequate contraction, Oxytocin infusion will start (five I.U. Oxytocin in 500 cc ringer I.V. drip) by titration method until complete regulation of uterine contractions.
      * Those with ruptured of membranes, the amniotic fluid color will be checked for any abnormalities and Oxytocin infusion will start (five I.U. Oxytocin in 500 cc ringer I.V. drip) by titration method until complete regulation of uterine contractions.
   2. If the contractions are adequate: No interference will be done.
6. Each participant will randomly take a prefilled syringe with two milliliters of the study medication solution (either Drotaverine Hydrochloride or saline). Each participant will take the selected syringe slowly intravenously over two minutes.
7. Partographic representation of labor and duration of first stage to determine the primary end point of the study "duration of 1st stage".
8. Cervical effacement and dilatation in addition to station and position of fetal head will be recorded every two hours by vaginal examination.
9. Reassessment after four hours of the first dose:

A) If poor progress: Initially, exclude C.P.D. & uterine inertia.

* If there is an obvious cause:

  * C.P.D.: Urgent C-section will be done.
  * Uterine inertia: adjust the dose of Oxytocin I.V drip via titration method until complete regulation of uterine contraction.
* If there is no obvious cause:

  * Another dose of the colorless solution will be given then reassessment after four hours, If no progress → re evaluation for final decision of mode of delivery.

B) If good progress: No interference will be done.

Outcome:

1. Primary outcomes:

   1. The duration of the active first stage of labor(Partographic representation for cervical effacement and dilatation will be plotted for each participant).
   2. Rate of cervical dilation (cm/h).
2. Secondary outcomes:

   1. Effect on pain by using visual analogue scale once before and one hour after injection of solution. VAS will be done at 30, 60 and 120 minutes of the drug administration.
   2. Mode of delivery.
   3. APGAR score less than 7 at 1 and 5 minutes.
   4. Maternal drug side effect will be recorded.

      Randomization and Blinding:

      Randomization will be achieved using a computer-generated randomization sequence. Allocation will be in a 1:1 ratio. Records of group allocation will be maintained by a resident physician "other than the researcher" whose responsibility will be randomization and drawing up the injection after dark sealing of the syringes with black opaque stickers to make the yellowish colored Drotaverine Hydrochloride (Do-Spa®) in-differentiable from the translucent saline solution.

      This house officer has no direct involvement in the intrapartum decision making. Drotaverine Hydrochloride and saline injections will have an identical appearance. The midwives, the clinicians staffing labor and delivery and the patients could not distinguish the placebo from the active drug. The randomization list will be held in a secure box on the labor ward to ensure concealment of the allocation of intervention from those recruiting participants.

      Data Collection:

      Maternal characteristics and labor information will be prospectively collected in a computerized database that will be maintained with daily chart review by the researcher to ensure accuracy and to minimize missing data The primary end-point of this study will be the duration of the first stage of labor.The first stage encompasses the onset of active labor to complete cervical dilatation.

      However, as women will be randomized at different dilatation levels, to allow meaningful comparison the dilatation rates (from administration of study drug

      o full dilatation) will be calculated and will be used as the primary outcome measure.

      Analysis:

      Data analysis and reporting will strictly follow the recommendation of CONSORT 2010 For each primary and secondary outcome, results for each group, and the estimated effect size and its precision (95% confidence interval).

      For binary outcomes, presentation of both absolute risk difference and relative (Risk Ratio) effect sizes will be reported.

      Ethical considerations

      IRB approval:

      The clinical research study will be conducted in accordance with the current IRB-approved clinical protocol; ICH GCP Guidelines; and relevant policies, requirements, and regulations of the Ain Shams University.

      Consent procedure:

      The investigator will make certain that an appropriate informed consent process is in place to ensure that potential research subjects, or their authorized representatives, are fully informed about the nature and objectives of the clinical study, the potential risks and benefits of study participation, and their rights as research subjects. The investigator will obtain written, signed informed consent of each subject, or the subject's authorized representative, prior to performing any study-specific procedures on the subject. The investigator will retain the original signed informed consent form.

      Subject confidentiality:

      All laboratory specimens, evaluation forms, reports, video recordings and other records that leave the site will not include unique personal data to maintain subject confidentiality.

      Funding: Internal funding by using the Hospital resources.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and less than 35 years.
* Primigravidae.
* Singleton pregnancy.
* Term gestation i.e., 37-42 weeks.
* Sure, reliable dates documented by ultrasound in the 1st half of pregnancy.
* Vertex presentation with occipito anterior position
* Regular uterine contractions at a rate of at least 3 to 4 contractions every 10 minutes, each contraction lasting for at least 40 seconds.
* Cervical dilatation of 3-5 cm.
* With or without rupture of membranes
* No evidence of maternal or fetal distress.

Exclusion Criteria:

* Cephalo-pelvic disproportion.
* Cervical surgery in the past or history of cervical injury.
* Patients on antihypertensive therapy.
* Known hypersensitivity to Drotaverine hydrochloride.
* If any other spasmolytic agent had been used within 48 hours.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Duration of the active first stage of labor | 12 hours

SECONDARY OUTCOMES:
Rate of cervical dilation (cm/h) | 12 hours
Effect on pain by using visual analogue scale | 12 hours
Mode of delivery | 12 hours
APGAR score less than 7 at 1 and 5 minutes | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ibrahem, MD, Study Director — Ain Shams University; Mohamed Ellaithy, MD, Study Chair — Ain Shams University
Locations (1):
- Labor at the delivery unit of Ain Shams Maternity Hospital, Al ‘Abbāsīyah, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Ibrahim MI, Ellaithy MI, Hussein AM, Nematallah MM, Allam HA, Abdelhamid AS, Harara RM, Riad AA, Rafaat TA. Measurement of maternal serum amyloid A as a novel marker of preterm birth. J Matern Fetal Neonatal Med. 2021 Aug;34(15):2467-2472. doi: 10.1080/14767058.2019.1668370. Epub 2019 Sep 25. PMID 31522581
- [Derived] Ibrahim MI, Alzeeniny HA, Ellaithy MI, Salama AH, Abdellatif MA. Drotaverine to improve progression of labor among nulliparous women. Int J Gynaecol Obstet. 2014 Feb;124(2):112-7. doi: 10.1016/j.ijgo.2013.08.013. Epub 2013 Nov 7. PMID 24299975
- See also: Ain Shams University — http://www.shams.edu.eg/